CLINICAL TRIAL: NCT04987164
Title: Observational Study Evaluating the Number of Symptomatic Cystitis-like Episodes and Urinary Comfort of Women Consuming Cranberry, Cinnamon and Probiotic Strain Extracts
Brief Title: Incidence of Cystitis in Women Consuming a Mixture of Cranberry, Cinnamon, Probiotics
Status: Completed | Type: Observational
Sponsor: CEN Biotech (Industry)
Collaborators: PiLeJe (Industry)
Responsible Party: Sponsor
Other Study IDs: C1671
Record Dates: First submitted 2021-07-19; First posted 2021-08-03 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Cystitis; Urinary Tract Infections
MeSH Terms: conditions — Cystitis; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Feminabiane CBU Consumers: Group of consumers of Feminabiane CBU : 2 tablets of Feminabiane CBU® every day, to be swallowed with a glass of water.
  Interventions: Dietary Supplement: Feminabiane CBU
- Control group: Control group of non consumers of Feminabiane CBU

INTERVENTIONS:
Dietary Supplement: Feminabiane CBU — EXTRACTS OF CRANBERRY, CINNAMON AND MICROBIOTIC STRAINS
  Groups: Feminabiane CBU Consumers

SUMMARY:
Cranberries are traditionally used for urinary comfort and prevention of urinary disorders of bacterial origin and despite an EFSA opinion invalidating the clinical efficacy of cranberries, its mechanism of action has been several times proposed by the scientific community: it would act by inhibiting the synthesis of P-fimbriae leading to a complete disappearance of these adhesins, and to bacterial-type deformation by lengthening of the cell body. Cinnamon and microbiotic strains could enhance this synergy.

This study aims to evaluate the effectiveness of a food supplement based on cranberry, cinnamon and microbiotic strains (Feminabiane CBU) on the symptoms of cystitis, urinary discomfort and the number of cystitis reported by women.

DETAILED DESCRIPTION:
Women who use or not the cranberry, cinnamon, and microbiotic blend are encouraged to complete a 6-month diary in which they report any urinary tract disorders they encounter.

ELIGIBILITY:
Inclusion Criteria:

* Having at least 2 symptomatic episodes of cystitis during the last 6 months including at least 1 episode confirmed as being bacterial cystitis (by an urine bacterial analysis or validated by a doctor (date of appointment, list of prescribed treatments) ;
* Whose symptomatic episodes of cystitis over the past 6 months have had a significant impact on quality of life / urinary comfort (ACSS QoL> 2);
* Having a smartphone compatible with the NURSTRIAL® data collection application;
* Not opposing the collection and processing of their personal data.

Exclusion Criteria:

* Presenting urinary discomfort with a severe impact on quality of life (ACSS QoL> 7) during the last 24 hours prior to inclusion;
* Pregnant, breastfeeding or planning to become pregnant during the study;
* Under antibiotic treatment (or during the last month preceding inclusion);
* Under food supplementation with prebiotics or probiotics or having stopped it less than a month before inclusion;
* Having had recourse to a prophylactic treatment (cranberry juice) 15 days before inclusion;
* Having had local estrogen therapy during the 3 months preceding inclusion;
* Diabetic;
* Presenting an immunosuppressive disease;
* Presenting pelvic floor abnormalities (Cystocele surgery, etc.);
* Presenting or having a history of kidney disease (including kidney stones, urinary tract abnormalities, pyelonephritis, kidney failure, kidney transplantation);
* For women consuming supplementation: known allergy to plants of the cranberry family or to one of the components of the products.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The first 80 women of the CEN Nutriment (Clinical Investigation Center) volunteer panel corresponding to the selection criteria and wishing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Occurence of symptomatic cystitis-like episodes | At week 24
  Number of symptomatic cystitis-like episodes reported by the subject self-assessed using the "typical" domain of the Acute Cystitis Symptom Score (ACCS) and defined by a score ranged between 6 to 18.

SECONDARY OUTCOMES:
Change of the quality of life related to urinary discomfort | At weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  ACCS "Quality of life" domain ranged between 0 (better) and 9 (worse)
Severity of urinary discomfort | Every day during each urinary symptoms (Week 0 to Week 24)
  Global ACCS score ranged between 0 (better) and 39 (worse)
Time-period without antibiotics | At week 24
  Measurement of the time interval between 2 antibiotic therapies if applicable
Mean time to onset of symptomatic episodes of the cystitis | At week 24
  Measurement of the time interval between 2 symptomatic episodes of the cystitis
Effect of blend consumption in preventing symptomatic episode of cystitis | At week 24
  Comparison of the rate of women blend users versus non-users who did not reported any symptomatic episode of cystitis as defined by a 0 score for the "typical" domain of the Acute Cystitis Symptom Score (ACCS).

OTHER OUTCOMES:
Assessing the remanent effect of the mix on total urinary tract disorders | At week 32
  Total number of urinary tract disorders reported by women, compared to the 0-24 week period
Assessing the remanent effect of the mix on the type urinary tract disorders | At week 32
  Rates of urinary tract disorders (cystitis and cystitis-like symptoms) reported by women, compared to the 0-24 week period
Satisfaction with the assessed mix | At month 1, 2, 3, 4, 5, 6
  Mean statisfaction score using a 5-point Likert scale: 1 means worse satisfaction and 5 means the best satisfaction.
  Very satisfied=1, Somewhat satisfied=2, Neither satisfied nor dissatisfied=3, Somewhat dissatisfied=4 and Very dissatisfied=5
Dietary supplementation ingestion observance | At weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Weekly number of food supplements not ingested in relation to the expected consumption
Gastrointestinal pain | At weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Visual analogic score assessing abdominal pain (0= no pain, 10= worse pain)
Gastrointestinal discomfort | At weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24
  Visual analogic score assessing bloating or flatulence (0= never, 10= always)
Assessing tolerance to the ingestion of food supplements | At week 24
  Total number encountered of adverse events (abdominal pain, bloating, constipation) and rates of this adverse events

CONTACTS AND LOCATIONS:
Overall Officials: JEAN-MARC BOHBOT, MD, Principal Investigator — Institut Fournier-PARIS
Locations (2):
- France (2):
  - CEN Nutriment, Dijon, Bourgogne-Franche-Comté
  - CEN Nutriment, Dijon, Burgundy

REFERENCES:
- [Derived] Ait Abdellah S, Leblanc A, Dauchet Q, Blondeau C, Bohbot JM. Effects of a supplement associating Lactobacillus strains and proanthocyanidin-rich plant extracts against recurrent uncomplicated, urinary tract infections: A prospective, controlled study. Investig Clin Urol. 2025 Jan;66(1):36-46. doi: 10.4111/icu.20240092. PMID 39791583